CLINICAL TRIAL: NCT00514436
Title: Case Management and Environmental Control in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ES 08711
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
Keywords: Asthma; children; low-income, underserved; Reduction in hospitalization
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Usual care consisted of referral back to primary care provider after index hospitalization
- Behavioral (Experimental): Asthma coaching, inperson contact followed by telephone contact
  Interventions: Behavioral: Asthma coaching

INTERVENTIONS:
Behavioral: Asthma coaching — Inperson contact followed by telephone with approach by issues raised by family
  Arms: Behavioral

SUMMARY:
Asthma among low-income, minority children remains a prime example of health disparities that are resistant to change. Controlled demonstrations of reductions in disproportionate hospital or emergency care are limited. We performed a controlled clinical trial of an "Asthma Coach" to reduce hospitalizations among low-income, African American children.

ELIGIBILITY:
Inclusion Criteria:

* 2-8 years of age
* Admitted to hospital for acute asthma
* African American ethnicity
* Medicaid coverage

Exclusion Criteria:

* Parent refusal to sign consent
* Living outside service area

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 1997-01; Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization | 2 years

SECONDARY OUTCOMES:
Emergency department visits | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Strunk, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States